CLINICAL TRIAL: NCT06937398
Title: Survey on Patient and Parental Perceptions of EEG-monitoring During Paediatric Anaesthesia Care
Status: Recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-2217
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Survey on Patient and Parental Perceptions of EEG-monitoring During Paediatric Anaesthesia Care
Keywords: EEG; Survey; Perception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study will include all parents of children aged one year and 16 yo and patients 12-16 yo: All parents of children 1-16 years old and patients 12-16 years old coming for elective surgery requiring GA at KK Women's and Children's Hospital will be invited to voluntarily participate in an electronic survey on Form SG.

SUMMARY:
Electroencephalographic (EEG) monitoring during general anaesthesia (GA) is not typically part of standard care during GA. The recent availability of non-invasive commercial EEG monitors for children has made EEG monitoring more popular. Several studies have shown that monitoring EEG while under GA allows customization and titration of GA. However, the usefulness of EEG monitoring in children have not been established. It is a relatively new technology for some and will involve additional costs. The investigators aim to understand the perceptions of participants regarding EEG monitoring during paediatric anaesthesia care by administering a survey before and after GA.

ELIGIBILITY:
Inclusion Criteria:

* All parents of children 1-16 years old and patients 12-16 years old coming for elective surgery requiring GA at KK Women's and Children's Hospital will be invited to voluntarily participate in an electronic survey on Form SG.

Exclusion Criteria:

* Parents and patients coming for emergency surgery will not be invited for the survey.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All parents of children 1-16 years old and patients 12-16 years old coming for elective surgery requiring GA at KK Women's and Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Survey on patient and parental perceptions of EEG-monitoring during paediatric anaesthesia care | May 2022 until September 2025
  Parents and patients completed the survey forms.

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Bong CL, Ho D, Allen JC, Lim GS, Tan HK, Broekman BFP, Fabila T, Reddy S, Koh WP, Swee-Kim Tan J, Meaney M, Rifkin-Graboi A. Early Neurodevelopmental Outcomes Following Exposure to General Anesthesia in Infancy: EGAIN, a Prospective Cohort Study. J Neurosurg Anesthesiol. 2023 Oct 1;35(4):394-405. doi: 10.1097/ANA.0000000000000857. Epub 2022 May 26. PMID 35613046